CLINICAL TRIAL: NCT04282746
Title: An Open-label, Single Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of Sublingually Administered (S)-Ketamine Oral Solution in Healthy Participants
Brief Title: A Study of Sublingually Administered (S)-Ketamine Oral Solution in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CR108751; 54135419EDI1002 (Other: Janssen Research & Development, LLC); 2019-004129-25 (EudraCT Number)
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JNJ-54135419 (Experimental): Participants will receive a single oral dose of JNJ-54135419-AAA oral solution for sublingual administration in 1 of 3 serial dose escalating cohorts in fasted conditions.
  Interventions: Drug: JNJ-54135419

INTERVENTIONS:
Drug: JNJ-54135419 — Single dose of JNJ-54135419 oral solution will be administered sublingually.
  Other Names: (S)-ketamine

SUMMARY:
The purpose of this study is to characterize the plasma pharmacokinetic (PK) profile following the single ascending dose (SAD) levels of an (S)-ketamine oral solution for sublingual administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20.0 and 28.0 kilogram per meter square kg/m^2 inclusive (BMI = weight/height^2) with a minimum weight of 60 kilogram (kg) and a maximum of 100 kg
* Participant must be healthy based on clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value that may lead to exclusion will be allowed once during the screening phase
* Non-smoker (not smoked for 3 months prior to screening)
* A woman must have a negative serum beta-human chorionic gonadotropin (beta-hCG) at screening and a negative urine pregnancy test prior to dosing on Day 1
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 1 month after the last study drug administration

Exclusion Criteria:

* Cardiac arrhythmias or other cardiac disease, hematological disease, hypertension, lipid abnormalities, respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, glaucoma, epilepsy or any other illness that the Investigator considers should exclude the participant
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies at screening visit
* Drinks, on average, more than 5 cups of tea/coffee/cocoa or 8 cans of cola per day
* Clinically significant acute illness within 7 days prior to study drug administration
* Donation of 1 or more units (approximately 450 milliliter [mL]) of blood or acute loss of an equivalent amount of blood within 90 days prior to study drug administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of (S)-ketamine | Predose, 1 minute (min), 3 min, 5 min, 10 min, 15 min, 30 min, 40 min, 1 hour (h), 1.5h, 2h, 3h, 4h, 6h, 8h, 12h and 24h postdose
  Observed plasma concentrations of (S)-ketamine will be reported.
Plasma Concentrations of Nor-(S)-ketamine | Predose, 1 minute (min), 3 min, 5 min, 10 min, 15 min, 30 min, 40 min, 1 hour (h), 1.5h, 2h, 3h, 4h, 6h, 8h, 12h and 24h postdose
  Observed plasma concentrations of nor-(S)-ketamine will be reported.

SECONDARY OUTCOMES:
Number of Participants with Vital Sign Abnormalities | Up to 4 Weeks
  Number of participants with vital signs (heart rate [HR], systolic blood pressure [SBP], diastolic blood pressure [DBP]) abnormalities will be reported.
Number of Participants with Adverse Events (AEs) | Up to 4 Weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Life Science Services, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency